CLINICAL TRIAL: NCT05901779
Title: Effect of Perioperative Probiotic Supplements on Postoperative Short-term Outcomes in Gastric Cancer Patients Receiving Neoadjuvant Chemotherapy: A Prospective, Randomized, Controlled, Multicenter Clinical Trial
Brief Title: Effect of Probiotic Supplements on Gastric Cancer Patients Receiving Neoadjuvant Chemotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Collaborators: Qilu Hospital of Shandong University (Other); Qianfoshan Hospital (Other); Shandong Provincial Hospital (Other Government); Yantai Yuhuangding Hospital (Other); Jining First People's Hospital (Other); Weifang Medical University (Other); Weifang People's Hospital (Other); Dongying People's Hospital (Other); Weihai Municipal Hospital (Other); Weihai Central Hospital (Other); Rizhao People's Hospital (Other); Liaocheng People's Hospital (Other); Qingdao Municipal Hospital (Other); The Second Hospital of Shandong University (Other); The People's Hospital of Jimo.Qingdao (Unknown); Binzhou People's Hospital (Other); Binzhou Medical University (Other); Jinan Central Hospital (Other); Shandong Cancer Hospital and Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GISSG2023-01
Record Dates: First submitted 2023-05-08; First posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Gastric Cancer; Neoadjuvant Chemotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Lacteol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic Group (Experimental): PG (probiotic group) patients received probiotic capsules containing Bifidobacterium longum, Lactobacillus acidophilus, and Enterococcus faecalis. The intervention begins from the completion of preoperative chemotherapy to the seventh day after surgery.
  Interventions: Drug: live combined Bifidobacteriun, Lactobacillus and Enterococcus capsules
- Control Group (No Intervention): CG (Control Group) patients receive blank control management.

INTERVENTIONS:
Drug: live combined Bifidobacteriun, Lactobacillus and Enterococcus capsules — Probiotics capsules containing Bifidobacterium longum, Lactobacillus acidophilus, and Enterococcus faecalis. Each capsule contained>10,000,000 colony-forming units (CFUs). This drug can treat endoxemia caused by imbalance of intestinal flora.
  Arms: Probiotic Group

SUMMARY:
Background: Surgery can significantly improve the prognosis of patients with gastric cancer. However, some patients are at a later stage at diagnosis and need to receive neoadjuvant chemotherapy (NACT). Previous studies have shown that NACT may lead to more postoperative complications. Probiotics have the potential to reduce postoperative complications and infections, but no large sample, multicentre, randomized clinical trials have been conducted in patients with gastric cancer receiving NACT. The aim of this multicentre randomized controlled trial was to investigate the effect of probiotics on postoperative infections and other short-term outcomes in patients with gastric cancer receiving NACT.

Methods/design: This study is a prospective, multicentre RCT. This experiment will consist of two groups - an experimental group and a control group - randomly divided in a 1:1 ratio. The experimental group will receive perioperative probiotic supplement and that of the control group will receive blank control management. An estimated 318 patients will be enrolled. The main endpoint for comparison is postoperative infections between the two groups.The experimental group patients received probiotic capsules containing Bifidobacterium longum, Lactobacillus acidophilus, and Enterococcus faecalis.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old
* male and female
* clinical stage was T3/4N+ evaluated by CT/MR/EUS at new diagnosis (before any anti-cancer treatment) , complete 2-4 cycles preoperative chemotherapy based on 5-FU (such as SOX, FLOX, ect.) at 3-6 weeks before surgery
* ASA grade was Ⅰ~Ⅲ
* radical minimal-invasive gastrectomy via laparoscope or DaVinci is judged as possible
* histologically confirmed gastric adenocarcinoma
* ECOG score is 0~1
* patients who provide a written informed consent before entering study screening

Exclusion Criteria:

* need emergency surgery due to performation and/or obstruction
* receive antibiotics and/or glucocorticoids within 14 days before surgery
* exist bacterial infection and/or autoimmune disease and/or IBD currently
* intolerance or allergic to probiotics
* upper abdominal surgery history
* use probiotics within 7 days before intervention, such as yogurt, ect.
* participate in other clinical trials currently
* severe mental illness
* can not participate in this trial due to severe illness of other organs evaluated by researchers, such as severe cardiac insufficiency (LVEF<30%, NYHA>Ⅱ, severe arrhythmia, congestive heart failure, myocardial infarction within 6 months), liver dysfunction (Child-Pugh C), renal dysfunction (need hemodialysis)
* need simultaneous surgery
* lactation or pregnancy
* refuse to participate in this trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
postoperative infectious complications | up tp 30 days after surgery
  The primary outcome was the incidence of postoperative infectious complications, which were defined as bacterial infections within 30 d after surgery. The diagnosis of infectious complications was based on fever (≥38°C), elevation of C-reactive protein (CRP), specific clinical symptoms of infection, and positive bacterial culture.

SECONDARY OUTCOMES:
postoperative recovery parameter | up tp 30 days after surgery
  time to first postoperative flatus and bowel movement; time to solid food tolerance; postoperative hospital stay;
postoperative death and readmission | up tp 30 days after surgery
  postoperative death and readmission within 30 days after surgery
duration of therapeutic antibiotic use | up tp 30 days after surgery
  duration of therapeutic antibiotic use measured as "day"
time to postoperative adjuvant chemotherapy | up tp 30 days after surgery
  durition from surgery to postoperative adjuvant chemotherapy.
European Organization for Reasearch and Treatment of Cancer Quality of Life Questionnare-Core 30 (EORTC QLQ-C30) (V3.0) | on postoperative day 30
  The European Organization for Reasearch and Treatment of Cancer Quality of Life Questionnare-Core 30, Higher scores for functional areas and general health indicate better functional status and quality of life, and higher scores for symptom areas indicate more symptoms or medical problems. The minimum value is 0 and maximum value is 100.
Postgastrectomy Syndrome Assessment Scale (PGSAS)-45 | on postoperative day 3, 5, and 30
  Higher score means more discomfort after gastrectomy. The minimum value is 0 and maximum value is 100
visual analogue scale | on postoperative day 1, 3 and 5
  from minimum 0 to maximun 10, higher score means more pain.
Leukocyte Count | Postoperative, on postoperative day 1, 3 and 5
  unit of measurement is "*10^9/L", recorded respectively according to measure time
percent of neutrophile granulocyte | Postoperative, on postoperative day 1, 3 and 5
  unit of measurement is "%", recorded respectively according to measure time
procalcitonin | Postoperative, on postoperative day 1, 3 and 5
  unit of measurement is "pg/ml", recorded respectively according to measure time
C-reactive protein | Postoperative, on postoperative day 1, 3 and 5
  unit of measurement is "mg/L", recorded respectively according to measure time
albumin | Postoperative, on postoperative day 1, 3 and 5
  unit of measurement is "*g/L", recorded respectively according to measure time
prealbumin | Postoperative, on postoperative day 1, 3 and 5
  unit of measurement is "mg/L", recorded respectively according to measure time
total bilirubin | Postoperative, on postoperative day 1, 3 and 5
  unit of measurement is "μmol/L", recorded respectively according to measure time

CONTACTS AND LOCATIONS:
Overall Officials: Yanbing Zhou, MD, Study Director — The Affiliated Hospital of Qingdao University
Locations (1):
- Department of Gastrointestinal Surgery, Qingdao University Affiliated Hospital, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Derived] Liu G, Cao S, Liu X, Tian Y, Yu W, Chai J, Li L, Wang X, Chu X, Duan Q, Qu J, Wang H, Zhang H, Wang X, Hui X, Yang D, Zhou S, Ding Y, Wang H, Zhou F, Hu B, Guo P, Jiang L, Zhang G, Pan Q, Zhou X, Zhou Y. Effect of perioperative probiotic supplements on the short-term clinical outcomes of patients undergoing laparoscopic or robotic radical gastrectomy after neoadjuvant chemotherapy: Study protocol for a multicenter randomized controlled trial (GISSG2023 - 01 Study). BMC Cancer. 2025 Apr 25;25(1):776. doi: 10.1186/s12885-025-14115-x. PMID 40281451